CLINICAL TRIAL: NCT06529276
Title: Augmented Reality Smart Glasses Technology for Immersive Learning in the Emergency Department (AGILE-1): a Pilot Randomised Controlled Study
Brief Title: Augmented Reality Smart Glasses Technology for Immersive Learning in the Emergency Department
Acronym: AGILE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lam Pui Kin, Clinical Associate Professor of Emergency Medicine, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AGILE1
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Augmented Reality
Keywords: Augmented reality; Smart glasses; Emergency airway management; Learning; Emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented reality (AR) clinical learning arm (Experimental): In the AR clinical learning arm, students will have one 3-hour session of AR clinical learning of emergency airway management. The PI will put on a HoloLens device and demonstrate endotracheal intubation using video laryngoscope (C-MAC®) and other AGPs, such as bag-valve-mask ventilation on a manikin in the resuscitation room. The students will be situated in another room and have a first-person view captured by the HoloLens during the demonstration.
  Interventions: Other: Augmented reality clinical learning
- Control clinical learning arm (Active Comparator): In the control arm, students will have one 3-hour regular session of bedside learning of emergency airway management. The PI will demonstrate endotracheal intubation using video laryngoscope (C-MAC®) and other AGPs, such as bag-valve-mask ventilation on a manikin in the resuscitation room in front of the students there.
  Interventions: Other: Control arm regular clinical learning

INTERVENTIONS:
Other: Augmented reality clinical learning — Clinical learning of emergency airway management including endotracheal intubation using video laryngoscope and other AGPs, such as bag-valve-mask ventilation, using augmented reality immersive learning technology.
  Arms: Augmented reality (AR) clinical learning arm
Other: Control arm regular clinical learning — Regular bedside learning of emergency airway management including endotracheal intubation using video laryngoscope and other AGPs, such as bag-valve-mask ventilation,
  Arms: Control clinical learning arm

SUMMARY:
The COVID-19 pandemic has disrupted traditional clinical teaching, depriving medical students of valuable clinical engagement with patients who required an aerosol-generating procedure (AGP) in the emergency department (ED). Because of the infection control restrictions, medical students are not allowed to enter resuscitation room where AGPs takes place, even in the aftermath of the pandemic.

The Microsoft HoloLens 2 is an augmented reality (AR) head-mounted device (HMD) which enables a single clinical teacher to facilitate real-time distant immersive learning by medical students on critically ill ED patients while insulating them from infection risks. Our team has successfully developed an AR HMD prototype based on HoloLens for clinical teaching and conducted 10 pilot teaching sessions. Overall, the audio-visual quality of the video-laryngoscope image captured by the HoloLens were rated satisfactorily by the students. Cybersickness symptoms such as dizziness, nausea, and eye strain were infrequent among the viewers.

The investigators conduct a pilot randomised controlled trial (RCT) which aims to evaluate the feasibility of conducting a full-scale RCT. The investigators collect data of the impact of AR learning and bedside learning on student knowledge gain, cognitive load, motivation and adverse effects. The investigators invite 33 Year 5 or 6 medical students to participate in this study during the Emergency Medicine Specialty Clerkship rotation at the Accident and Emergency Department (A&E) of Queen Mary Hospital (QMH). Consented medical students are randomly assigned in clusters based on their existing student group assignment (around 10 students per each small group) in a 1:1 to two arms: AR clinical learning arm and the control arm (bedside clinical learning).

Randomisation is performed by a research assistant not directly involved in the study using sequentially numbered opaque, sealed envelopes. Given the first-person perspective through the HoloLens, it is not possible to blind the medical students.

To standardise the teaching content of all study sessions, all such sessions are delivered by the principal investigator (PI) of this study during the study period and the pre-reading materials are the same for both groups. The PI will demonstrate endotracheal intubation using video laryngoscope and other AGPs on a manikin in the resuscitation room.

ELIGIBILITY:
Inclusion Criteria:

* Year 5 or 6 medical students during the Emergency Medicine Specialty Clerkship

Exclusion Criteria:

* refusal to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Knowledge gain (in full-scale RCT) | Immediately after the AR/control learning session
  Knowledge gain measured with pre- and post-AR/control session knowledge tests, which consist of 20 multiple choice questions on emergency airway management

SECONDARY OUTCOMES:
Student domain interest | Immediately after the AR/control learning session
  Student interest in emergency airway management assessed with 3 questions (e.g. "I know a lot about emergency airway management.") with responses captured using 100 mm visual analogue scales. To each of these questions, the answer ranges from 0 to 100 on a VAS where 0 is complete disagreement and 100 is perfect agreement with the statement.
Student opinion on the learning method | Immediately after the AR/control learning session
  Student opinion on the learning method assessed with 5 questions (e.g. "The learning method is highly effective for me to learn about emergency airway management.") with responses captured using 100 mm visual analogue scales. To each of these questions, the answer ranges from 0 to 100 on a VAS where 0 is complete disagreement and 100 is perfect agreement with the statement.
Student perceived motivation | Immediately after the AR/control learning session
  Student perceived motivation assessed with 4 questions (e.g. "The quality of the clinical session helped to hold my attention.") with responses captured using 100 mm visual analogue scales. To each of these questions, the answer ranges from 0 to 100 on a VAS where 0 is complete disagreement and 100 is perfect agreement with the statement.
Self-efficacy | Immediately after the AR/control learning session
  Student self-efficacy assessed with 5 questions (e.g."I am confident that I will be able to master the skills taught in this clinical session.") with responses captured using 100 mm visual analogue scales. To each of these questions, the answer ranges from 0 to 100 on a VAS where 0 is complete disagreement and 100 is perfect agreement with the statement.
Student cognitive load | Immediately after the AR/control learning session
  Student cognitive load assessed with 7 questions (e.g. "For this clinical session, many things needed to be kept in mind simultaneously.") with responses captured using 100 mm visual analogue scales. To each of these questions, the answer ranges from 0 to 100 on a VAS where 0 is complete disagreement and 100 is perfect agreement with the statement.
Adverse health effects | Immediately after the AR/control learning session
  Adverse health effects during the learning session such as symptoms of cybersickness assessed including dizziness and nausea using 7-point Likert scale, with higher numerical scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Rex Pui Kin Lam, MBBS, FHKCEM, Principal Investigator — Rex Pui Kin Lam
Locations (1):
- Accident and Emergency Department, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Data could be shared with other researchers upon reasonable requests and after additional approval by the institutional review board.